CLINICAL TRIAL: NCT03201432
Title: A Randomized Trial for Treatment of Symptomatic Extracranial Vertebral Artery Stenosis: Drug Eluting Stents Versus Bare Metal Stents
Brief Title: Drug Eluting Stents Versus Bare Metal Stents for Treatment of Symptomatic Extracranial Vertebral Artery Stenosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiongjing Jiang (Other)
Collaborators: Yinyi(Liaoning) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-ZX15
Record Dates: First submitted 2016-03-04; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Stroke; Vertebral Artery Stenosis
Keywords: Vertebral Artery Stenosis; Ischemic Stroke; Stent
MeSH Terms: conditions — Ischemic Stroke; Vertebrobasilar Insufficiency | interventions — Drug-Eluting Stents

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bare metal stent (BES) group (Other): Percutaneous vertebral artery stenting using bare metal stents (Boston Scientific：Express SD) in patients randomized to BES group
  Interventions: Device: Bare metal stent (BES)
- Drug eluting stent (DES) group (Experimental): Percutaneous vertebral artery stenting using drug eluting stents (Liaoning Biomedical Materials R&D Center Co., Ltd. ：YINYI) in patients randomized to DES group
  Interventions: Device: Drug eluting stent (DES)

INTERVENTIONS:
Device: Drug eluting stent (DES) — Polymer-free paclitaxel eluting stents
  Other Names: YINYI (Liaoning Biomedical Materials R&D Center Co., Ltd.)
  Arms: Drug eluting stent (DES) group
Device: Bare metal stent (BES) — Bare metal stent
  Other Names: Express SD (Bosten Scientific)
  Arms: Bare metal stent (BES) group

SUMMARY:
Stroke is one of the important causes of disability and death in the world, in which more than half were ischemic strokes. About 1/4 of the ischemic stroke occurred in the vertebral basilar artery system, especially when in the presence of extracranial proximal vertebral artery stenosis. Vertebral artery stenting is a minimally invasive method for the reconstruction of vertebral artery stenosis and the early clinical studies showed that it was feasible, safe and effective, but the high rate of restenosis has become a bottleneck restricting its development. Previous systematic review had suggested that the drug eluting stent might reduce the incidence of restenosis of vertebral artery. However, prospective randomized controlled trials comparing the efficacy of bare metal stents and drug eluting stents on the prevention of restenosis remains absent.

DETAILED DESCRIPTION:
60 patients were randomly assigned into DES and BES group to compare the safety and efficacy in the treatment of symptomatic extracranial vertebral artery stenosis with drug eluting stents (YINYI) and bare metal stents (Express SD), especially the stent restenosis rate after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic posterior circulation ischemia（Vertebral basilar artery system TIA or non-disabling ischemic stroke）result from the stenosis in the extracranial proximal vertebral artery stenosis.
* Atherosclerotic extracranial proximal vertebral artery stenosis demonstrated by angiography(any of the following): 1) bilateral vertebral artery stenosis ≥70%, or vertebral artery stenosis ≥70% concomitant occlusion of contralateral vertebral artery; 2) superior lateral vertebral artery stenosis ≥70%; 3) non-superior lateral vertebral artery stenosis ≥50%, but the vertebral artery was directly extended to the posterior inferior cerebellar artery on this side and symptoms were related to insufficiency of the ipsilateral posterior inferior cerebellar artery.

Exclusion Criteria:

* 1) lesions characteristics (such as diffuse lesions) which was not suitable for interventional treatment, or unstable condition that cannot tolerate the interventional therapy;
* 2) vertebral artery stenosis caused by non atherosclerosis disease: Takayasu arteritis or other diseases;
* 3) severe stroke within 3 months;
* 4) contraindicated using contrast agents: such as chronic renal insufficiency or had serious contrast agents allergy history;
* 5) malignant tumor;
* 6) with Alzheimer's disease or mental illness previously or currently ;
* 7) patients or family members refuse the operation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Stent restenosis rate 6 months after stenting | 6 months

SECONDARY OUTCOMES:
Stent restenosis rate 3 months after stenting | 3 months
Stent restenosis rate 12 months after stenting | 12 months
  measured by ultrasound
The incidence of cardiovascular events (stroke, TIA, Miocardial infarction and death) 6 months after stenting | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, M.D., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: No